CLINICAL TRIAL: NCT01112137
Title: Phase IV Study of the Effects of Clopidogrel on Soluble CD40 Ligand, Endothelial Function and Blood Pressure
Brief Title: Effects of Clopidogrel on Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Dirk Taubert, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NLN5031
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Blood Pressure; Endothelial Function; Platelet Function
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hypertensive individuals: clopidogrel (600 mg, bolus) (Experimental)
  Interventions: Drug: Clopidogrel
- Hypertensive individuals: clopidogrel (75 mg daily) (Experimental)
  Interventions: Drug: Clopidogrel
- Normotensive individuals: clopidogrel (600 mg, bolus) (Active Comparator)
  Interventions: Drug: Clopidogrel
- Normotensive individuals: clopidogrel (75 mg, daily) (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel
  Arms: Hypertensive individuals: clopidogrel (600 mg, bolus)
Drug: Clopidogrel
  Arms: Hypertensive individuals: clopidogrel (75 mg daily)
Drug: Clopidogrel
  Arms: Normotensive individuals: clopidogrel (600 mg, bolus)
Drug: Clopidogrel
  Arms: Normotensive individuals: clopidogrel (75 mg, daily)

SUMMARY:
Context: Soluble CD40 ligand (sCD40L) released from activated platelets induces inflammatory transformation of the vascular endothelium and is an independent predictor of cardiovascular events. Arterial hypertension is associated with platelet activation, increased sCD40L levels and endothelial dysfunction suggesting that inhibition of platelet-derived sCD40L release may improve endothelial function and lower blood pressure (BP).

Objective: To determine the effects of clopidogrel on sCD40L, endothelial function and BP.

Design: Randomized, controlled, investigator-blinded, parallel-group, 2-phase trial in patients with coronary artery disease and essential arterial hypertension and those without hypertension.

Intervention: Participants receive a single 600-mg clopidogrel loading dose (phase I) followed by a daily 75-mg clopidogrel maintenance dose over 28 days (phase II).

Outcome Measures: Primary outcome measure is the change in BP from baseline. Secondary outcome measures are changes in biomarkers of platelet and endothelial function and their correlation with BP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease (CAD) and a clinical presentation of stable angina pectoris or acute coronary syndrome who had undergone percutaneous coronary intervention (PCI) with stent implantation
* 5-year history of essential arterial hypertension with a systolic BP between 140 and 170 mmHg or no hypertension (systolic BP <140mg Hg and diastolic BP <90 mmHg)
* treatment with clopidogrel (75 mg per day) for 6 to 12 months after PCI
* continuous use of aspirin (100 mg per day)
* no change in drug therapy within 3 months prestudy

Exclusion Criteria:

* stent thrombosis or another ischemic cardiovascular event following PCI
* use of other antiplatelet drugs or anticoagulants within 3 months prestudy
* surgery within 3 months prestudy
* arrhythmia
* valvular heart disease
* hematologic disorder
* severe renal disorder
* severe hepatic disorder
* chronic inflammatory disorder
* autoimmune disorder
* acute or chronic infection
* active malignancy
* a body-mass index below 18.5 or above 40 kg/m2
* nonadherence to therapy
* nonattendance to control visits

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
blood pressure

SECONDARY OUTCOMES:
markers of platelet and endothelial function

CONTACTS AND LOCATIONS:
Locations (2):
- University of Cologne, Cologne, Germany
- St Antonius Hospital Nieuwegein, Nieuwegein, Netherlands

REFERENCES:
- [Background] Heeschen C, Dimmeler S, Hamm CW, van den Brand MJ, Boersma E, Zeiher AM, Simoons ML; CAPTURE Study Investigators. Soluble CD40 ligand in acute coronary syndromes. N Engl J Med. 2003 Mar 20;348(12):1104-11. doi: 10.1056/NEJMoa022600. PMID 12646667
- [Background] Heitzer T, Rudolph V, Schwedhelm E, Karstens M, Sydow K, Ortak M, Tschentscher P, Meinertz T, Boger R, Baldus S. Clopidogrel improves systemic endothelial nitric oxide bioavailability in patients with coronary artery disease: evidence for antioxidant and antiinflammatory effects. Arterioscler Thromb Vasc Biol. 2006 Jul;26(7):1648-52. doi: 10.1161/01.ATV.0000225288.74170.dc. Epub 2006 May 4. PMID 16675725
- [Background] Henn V, Slupsky JR, Grafe M, Anagnostopoulos I, Forster R, Muller-Berghaus G, Kroczek RA. CD40 ligand on activated platelets triggers an inflammatory reaction of endothelial cells. Nature. 1998 Feb 5;391(6667):591-4. doi: 10.1038/35393. PMID 9468137
- [Background] Chen C, Chai H, Wang X, Jiang J, Jamaluddin MS, Liao D, Zhang Y, Wang H, Bharadwaj U, Zhang S, Li M, Lin P, Yao Q. Soluble CD40 ligand induces endothelial dysfunction in human and porcine coronary artery endothelial cells. Blood. 2008 Oct 15;112(8):3205-16. doi: 10.1182/blood-2008-03-143479. Epub 2008 Jul 24. PMID 18658029